CLINICAL TRIAL: NCT04389203
Title: Pregnancy Rate After Laparoscopic Unilateral Tubal Disconnection
Brief Title: Pregnancy Rate After Unilateral Tubal Disconnection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRAUTD
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Rate
Keywords: pregnancy rate; Lasparosocpy; Unilateral tubal disconnection; Intracytoplasmic sperm injection
MeSH Terms: interventions — Pregnancy; Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: Unilateral tubal disconnection and spontaneous pregnancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Unilateral tubal disconnection and waiting for pregnancy for 2 years after laparoscopy
  Interventions: Procedure: Unilateral tubal disconnection + Spontaneous follow up for pregnancy
- Control group (Experimental): Unilateral tubal disconnection and ICSI
  Interventions: Procedure: Unilateral tubal disconnection + ICSI

INTERVENTIONS:
Procedure: Unilateral tubal disconnection + Spontaneous follow up for pregnancy — Unilateral tubal disconnection + Spontaneous follow up for pregnancy
  Arms: Study group
Procedure: Unilateral tubal disconnection + ICSI — Unilateral tubal disconnection + ICSI
  Arms: Control group

SUMMARY:
Unilateral disconnection of one tube that had hydrosalpinx

DETAILED DESCRIPTION:
In cases suffering from infertility and all other factors were normal except hysterosalpingogram that showed hydrosalpinx.

We either did intracytoplasmic sperm injection (ICSI) in one group and spontaneous follow up for 2 years after laparoscopy Pregnancy rate in both groups was assessed

ELIGIBILITY:
Inclusion Criteria:

* infertile women either primary or secondary Hydrosalpinx

Exclusion Criteria:

* other factors of infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 2 years
  Number of pregnant women after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Adel Elgergawy, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
When we finish the results
Supporting Information: Study Protocol
Time Frame: 6 months